CLINICAL TRIAL: NCT00136032
Title: Gender-Specific Effects of Physiologic GH Administration on Cardiovascular Risk Factors in Women With Growth Hormone Deficiency
Brief Title: Growth Hormone Administration and Its Effects on Cardiovascular Risk Factors in Growth Hormone Deficient Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Anne Klibanski, MD, Massachusetts General Hospital / Harvard Medical School
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2001p-001761
Record Dates: First submitted 2005-08-24; First posted 2005-08-26 (Estimated); Last update posted 2008-02-18 (Estimated); Status verified 2008-02

CONDITIONS: Growth Hormone Deficiency
Keywords: Growth Hormone; Cardiovascular risk; Pituitary; Hypothalamic; GH Deficiency; Pituitary Tumor; Pituitary Disease
MeSH Terms: conditions — Dwarfism, Pituitary; Pituitary Diseases; Pituitary Neoplasms | interventions — Human Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Somatropin
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Somatropin — Stratified based on age and estrogen status from 3 to 6 mcg/kg/day
  Other Names: Genotropin
  Arms: 1
Drug: Placebo — Dosage based on age and estrogen status ranging from 3 to 6 mcg/kg/day
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate the effects of growth hormone replacement on women with growth hormone deficiency. Growth hormone deficiency means the body no longer produces growth hormone due to a tumor or some kind of disease of the brain in an area called the pituitary/hypothalamic region. This is the area of the brain where growth hormone is normally produced. We, the researchers at Massachusetts General Hospital, will establish the effects of growth hormone replacement on cardiovascular parameters (laboratory tests, the flexibility of the arteries, changes in heart rate) in women with growth hormone deficiency. Our goal is to see if this therapy:

* has effects on women's cardiovascular risk markers (special blood tests which indicate how healthy the heart and arteries are)
* has effects on women's types and levels of various substances circulating in their blood
* in women affects the stiffness of their arteries and heart rate variability in parallel with changes in cardiovascular risk markers
* has different effects depending on whether women are pre or post menopausal.

Participation in this study is expected to last approximately 12 months.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the gender specific effects of physiologic Growth Hormone (GH) replacement in women with GH deficiency on the basis of pituitary/hypothalamic region tumors, radiation, or surgery on cardiovascular risk markers and arterial distensibility. Cardiovascular mortality in growth hormone (GH) deficient adults has been shown to be increased in a number of retrospective studies. Increased arterial intima-media thickness, increased prevalence of atherosclerotic plaques and endothelial dysfunction have been reported in growth hormone deficient adults both in childhood and adulthood onset forms.

The growth hormone deficiency (GHD) syndrome is associated with a cluster of cardiovascular-risk factors such as central adiposity, increased visceral fat, insulin resistance, dyslipoproteinemia and decreased plasma fibrinolytic activity. GH administration has effects on a number of these factors, but it is unknown which mechanisms are implicated in GH action on the process of atherosclerosis. In addition to alterations in atherosclerotic markers, abnormalities in cardiac function and structure have been reported among patients with GHD possibly contributing to the increased cardiovascular mortality. In addition, GHD is associated with cardiac autonomic dysfunction that may also contribute to cardiovascular mortality and improves with GH replacement therapy.

The vast majority of studies have focused primarily on men and the gender-specific effects of GH replacement on cardiovascular risk factors remain unknown. In addition to being of interest in terms of understanding the physiologic effects of GH therapy, there are important therapeutic implications regarding data in women. Cardiovascular disease is the leading cause of mortality in women. Effects of GH replacement on bone density may be less pronounced in women and because specific GH effects on cardiovascular risk factors in women are unknown, many adult women with GHD are untreated.

Long-term GH treatment decreases total body fat including visceral fat. Decreases in central fat as assessed by waist to hip ratio have been reported in some studies, but not in others. Administration of GH causes insulin resistance acutely but long-term therapy may restore glucose sensitivity. GH treatment increases lipoprotein (a) (Lp (a)) levels but its effects on other lipoproteins are still controversial. Some studies have reported decreases in LDL cholesterol with or without increases in HDL cholesterol with GH administration, while others have not. Twelve months of GH replacement improves left ventricular mass and cardiac performance in young adults with GHD. Key factors likely involved in the discrepant findings include heterogeneity of patients studied in terms of age of onset of the GH deficiency (childhood versus adulthood), gender, severity of GHD and methodologic issues such as dose and duration of GH administration. In addition, many of the studies have no control period.

Inflammation plays a central role in the pathophysiology of atherosclerosis. Each atherosclerotic lesion represents a different stage of a chronic inflammatory process in the arterial wall and different markers along the inflammatory cascade have been reported to predict cardiovascular risk [34]. Among those, high-sensitivity testing for C-reactive protein (CRP) is one of the best validated. Several prospective studies support a strong link between levels of CRP and future risk of coronary events. CRP adds considerable value to the total and HDL cholesterol measurement in the prediction of cardiovascular risk. Other distal indicators of inflammation such as serum-amyloid polypeptide A (SAA) likewise predict coronary risk. These distal markers reflect the consequences of elevated proinflammatory cytokines like interleukin-6 (IL-6). GH is known to have important immunomodulatory effects. We therefore hypothesized that the effects of GH on the process of atherosclerosis might be mediated through the cytokine-inflammatory pathway. We have recently investigated the effects of physiologic GH replacement in cardiovascular risk markers in men with GHD. In this study we found that CRP and IL-6 levels decreased in GH treated men compared to controls despite no significant change in serum lipid levels. We also recently have investigated levels of inflammatory markers in women with hypopituitarism compared with healthy controls. We found that women with hypopituitarism have increased levels of IL-6 and CRP suggesting that chronic inflammation may be involved in the pathogenesis of atherosclerosis in this population. It will be critical to determine whether physiologic GH replacement has beneficial effects in women, and whether these effects are influenced by estrogen.

We will investigate the effect of long-term physiologic GH administration on IL-6, CRP, SAA as well as other classic cardiovascular risk factors in women with GHD in a randomized, placebo-controlled study. In addition, we will evaluate structural/function correlates in women by measuring arterial wall distensibility and heart rate variability in parallel with cardiovascular risk markers.

We will establish the gender-specific effects of physiologic GH replacement on cardiovascular risk in women with GHD by investigating whether this therapy:

1. has gender-specific effects on cardiovascular risk markers
2. has gender-specific effects on lipid profiles
3. alters heart rate variability and arterial distensibility in parallel with changes in cardiovascular risk markers
4. has different effects depending upon gonadal status

ELIGIBILITY:
Inclusion Criteria:

* GH deficiency due to pituitary or hypothalamic tumors or disease affecting this area. Subjects will have been treated with medication, surgery, radiation, or a combination of these. GH deficiency will be defined as a peak plasma GH of less than 5 ng/ml in response to insulin tolerance testing or growth hormone releasing hormone (GHRH) plus arginine stimulation test. In subjects with suspected hypothalamic dysfunction the arginine plus L-dopa stimulation test may be used, with a cutoff of 1.7 ng/ml for diagnosis of GH deficiency. Partial GH deficiency will be defined as a GH peak of 5 to 9 ng/ml (inclusive) during insulin tolerance testing or GHRH plus arginine testing.
* GH deficiency will also be diagnosed if insulin-like growth factor-I (IGF-I) levels are below 2 standard deviations for the age-sex normal range in a patient with at least two documented hormone deficiencies.
* Subjects must have evidence of a stable pituitary mass (for at least 12 months) if there is a history of a tumor except in the case of ACTH-producing microadenomas, where no follow-up imaging is required after cure.
* Subjects age 40 and over must have a screening mammogram if they have not already had one within one year prior to their baseline visit

Exclusion Criteria:

* Active Cushing's disease within 1 year
* History of acromegaly
* Untreated thyroid or adrenal insufficiency. Subjects on replacement therapy must be stable for at least 3 months prior to entry into the study.
* History of malignancy except for skin cancer and except for childhood solid malignancy with documented cure for > 10 years prior to starting the study
* Hemoglobin <10.0 gm/dl
* Hepatic or renal disease (SGPT/SGOT > 3x upper limit of normal (ULN) or creatinine levels >2.5 mg/dl)
* Congestive heart failure (CHF) (New York Heart Association's classification system Class II-IV CHF will be excluded)
* History of unstable cardiovascular disease (coronary artery or cerebrovascular disease) or symptoms within one year prior to entry into the study
* Diabetes mellitus
* Pregnancy or nursing
* Active carpal tunnel syndrome

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2002-01; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Gender specific effects on cardiovascular risk markers | baseline, 1, 3, 6, 7, 9, and 12 months

SECONDARY OUTCOMES:
Heart Rate Variability | baseline, 3, 6, 9, and 12 months
Quality of Life | baseline, 1, 3, 6, 7, 9, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anne Klibanski, M.D, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Rosen T, Bengtsson BA. Premature mortality due to cardiovascular disease in hypopituitarism. Lancet. 1990 Aug 4;336(8710):285-8. doi: 10.1016/0140-6736(90)91812-o. PMID 1973979
- [Background] Bulow B, Hagmar L, Eskilsson J, Erfurth EM. Hypopituitary females have a high incidence of cardiovascular morbidity and an increased prevalence of cardiovascular risk factors. J Clin Endocrinol Metab. 2000 Feb;85(2):574-84. doi: 10.1210/jcem.85.2.6346. PMID 10690858
- [Background] Wuster C, Slenczka E, Ziegler R. [Increased prevalence of osteoporosis and arteriosclerosis in conventionally substituted anterior pituitary insufficiency: need for additional growth hormone substitution?]. Klin Wochenschr. 1991 Oct 18;69(16):769-73. doi: 10.1007/BF01797616. German. PMID 1762381
- [Background] Tomlinson JW, Holden N, Hills RK, Wheatley K, Clayton RN, Bates AS, Sheppard MC, Stewart PM. Association between premature mortality and hypopituitarism. West Midlands Prospective Hypopituitary Study Group. Lancet. 2001 Feb 10;357(9254):425-31. doi: 10.1016/s0140-6736(00)04006-x. PMID 11273062
- [Background] Markussis V, Beshyah SA, Fisher C, Sharp P, Nicolaides AN, Johnston DG. Detection of premature atherosclerosis by high-resolution ultrasonography in symptom-free hypopituitary adults. Lancet. 1992 Nov 14;340(8829):1188-92. doi: 10.1016/0140-6736(92)92892-j. PMID 1359261
- [Background] Pfeifer M, Verhovec R, Zizek B, Prezelj J, Poredos P, Clayton RN. Growth hormone (GH) treatment reverses early atherosclerotic changes in GH-deficient adults. J Clin Endocrinol Metab. 1999 Feb;84(2):453-7. doi: 10.1210/jcem.84.2.5456. PMID 10022400
- [Background] Evans LM, Davies JS, Goodfellow J, Rees JA, Scanlon MF. Endothelial dysfunction in hypopituitary adults with growth hormone deficiency. Clin Endocrinol (Oxf). 1999 Apr;50(4):457-64. doi: 10.1046/j.1365-2265.1999.00671.x. PMID 10468904
- [Background] Capaldo B, Patti L, Oliviero U, Longobardi S, Pardo F, Vitale F, Fazio S, Di Rella F, Biondi B, Lombardi G, Sacca L. Increased arterial intima-media thickness in childhood-onset growth hormone deficiency. J Clin Endocrinol Metab. 1997 May;82(5):1378-81. doi: 10.1210/jcem.82.5.3951. PMID 9141519
- [Background] Cuneo RC, Salomon F, McGauley GA, Sonksen PH. The growth hormone deficiency syndrome in adults. Clin Endocrinol (Oxf). 1992 Nov;37(5):387-97. doi: 10.1111/j.1365-2265.1992.tb02347.x. No abstract available. PMID 1486686
- [Background] De Boer H, Blok GJ, Voerman HJ, De Vries PM, van der Veen EA. Body composition in adult growth hormone-deficient men, assessed by anthropometry and bioimpedance analysis. J Clin Endocrinol Metab. 1992 Sep;75(3):833-7. doi: 10.1210/jcem.75.3.1517374.
- [Background] Binnerts A, Deurenberg P, Swart GR, Wilson JH, Lamberts SW. Body composition in growth hormone-deficient adults. Am J Clin Nutr. 1992 May;55(5):918-23. doi: 10.1093/ajcn/55.5.918. PMID 1570798
- [Background] Weaver JU, Monson JP, Noonan K, John WG, Edwards A, Evans KA, Cunningham J. The effect of low dose recombinant human growth hormone replacement on regional fat distribution, insulin sensitivity, and cardiovascular risk factors in hypopituitary adults. J Clin Endocrinol Metab. 1995 Jan;80(1):153-9. doi: 10.1210/jcem.80.1.7829604.
- [Background] Johansson JO, Fowelin J, Landin K, Lager I, Bengtsson BA. Growth hormone-deficient adults are insulin-resistant. Metabolism. 1995 Sep;44(9):1126-9. doi: 10.1016/0026-0495(95)90004-7. PMID 7666785
- [Background] Rosen T, Eden S, Larson G, Wilhelmsen L, Bengtsson BA. Cardiovascular risk factors in adult patients with growth hormone deficiency. Acta Endocrinol (Copenh). 1993 Sep;129(3):195-200. doi: 10.1530/acta.0.1290195. PMID 8212983
- [Background] Johansson JO, Landin K, Tengborn L, Rosen T, Bengtsson BA. High fibrinogen and plasminogen activator inhibitor activity in growth hormone-deficient adults. Arterioscler Thromb. 1994 Mar;14(3):434-7. doi: 10.1161/01.atv.14.3.434. PMID 8123648
- [Background] Shahi M, Beshyah SA, Hackett D, Sharp PS, Johnston DG, Foale RA. Myocardial dysfunction in treated adult hypopituitarism: a possible explanation for increased cardiovascular mortality. Br Heart J. 1992 Jan;67(1):92-6. doi: 10.1136/hrt.67.1.92. PMID 1739534
- [Background] Longobardi S, Cuocolo A, Merola B, Di Rella F, Colao A, Nicolai E, Cardei S, Salvatore M, Lombardi G. Left ventricular function in young adults with childhood and adulthood onset growth hormone deficiency. Clin Endocrinol (Oxf). 1998 Feb;48(2):137-43. doi: 10.1046/j.1365-2265.1998.00281.x. PMID 9579223
- [Background] Leong KS, Mann P, Wallymahmed M, MacFarlane IA, Wilding JP. Abnormal heart rate variability in adults with growth hormone deficiency. J Clin Endocrinol Metab. 2000 Feb;85(2):628-33. doi: 10.1210/jcem.85.2.6396. PMID 10690867
- [Background] Cuneo RC, Judd S, Wallace JD, Perry-Keene D, Burger H, Lim-Tio S, Strauss B, Stockigt J, Topliss D, Alford F, Hew L, Bode H, Conway A, Handelsman D, Dunn S, Boyages S, Cheung NW, Hurley D. The Australian Multicenter Trial of Growth Hormone (GH) Treatment in GH-Deficient Adults. J Clin Endocrinol Metab. 1998 Jan;83(1):107-16. doi: 10.1210/jcem.83.1.4482. PMID 9435425
- [Background] Baum HB, Biller BM, Finkelstein JS, Cannistraro KB, Oppenhein DS, Schoenfeld DA, Michel TH, Wittink H, Klibanski A. Effects of physiologic growth hormone therapy on bone density and body composition in patients with adult-onset growth hormone deficiency. A randomized, placebo-controlled trial. Ann Intern Med. 1996 Dec 1;125(11):883-90. doi: 10.7326/0003-4819-125-11-199612010-00003. PMID 8967668
- [Background] Bengtsson BA, Eden S, Lonn L, Kvist H, Stokland A, Lindstedt G, Bosaeus I, Tolli J, Sjostrom L, Isaksson OG. Treatment of adults with growth hormone (GH) deficiency with recombinant human GH. J Clin Endocrinol Metab. 1993 Feb;76(2):309-17. doi: 10.1210/jcem.76.2.8432773.
- [Background] Jorgensen JO, Pedersen SA, Thuesen L, Jorgensen J, Ingemann-Hansen T, Skakkebaek NE, Christiansen JS. Beneficial effects of growth hormone treatment in GH-deficient adults. Lancet. 1989 Jun 3;1(8649):1221-5. doi: 10.1016/s0140-6736(89)92328-3. PMID 2566779
- [Background] Salomon F, Cuneo RC, Hesp R, Sonksen PH. The effects of treatment with recombinant human growth hormone on body composition and metabolism in adults with growth hormone deficiency. N Engl J Med. 1989 Dec 28;321(26):1797-803. doi: 10.1056/NEJM198912283212605. PMID 2687691
- [Background] Florkowski CM, Collier GR, Zimmet PZ, Livesey JH, Espiner EA, Donald RA. Low-dose growth hormone replacement lowers plasma leptin and fat stores without affecting body mass index in adults with growth hormone deficiency. Clin Endocrinol (Oxf). 1996 Dec;45(6):769-73. doi: 10.1046/j.1365-2265.1996.830895.x. PMID 9039344
- [Background] Whitehead HM, Boreham C, McIlrath EM, Sheridan B, Kennedy L, Atkinson AB, Hadden DR. Growth hormone treatment of adults with growth hormone deficiency: results of a 13-month placebo controlled cross-over study. Clin Endocrinol (Oxf). 1992 Jan;36(1):45-52. doi: 10.1111/j.1365-2265.1992.tb02901.x. PMID 1559299
- [Background] Fowelin J, Attvall S, Lager I, Bengtsson BA. Effects of treatment with recombinant human growth hormone on insulin sensitivity and glucose metabolism in adults with growth hormone deficiency. Metabolism. 1993 Nov;42(11):1443-7. doi: 10.1016/0026-0495(93)90197-v. PMID 8231841
- [Background] Nolte W, Radisch C, Armstrong VW, Hufner M, von zur Muhlen A. The effect of recombinant human GH replacement therapy on lipoprotein(a) and other lipid parameters in adults with acquired GH deficiency: results of a double-blind and placebo-controlled trial. Eur J Endocrinol. 1997 Nov;137(5):459-66. doi: 10.1530/eje.0.1370459. PMID 9405024
- [Background] Beshyah SA, Henderson A, Niththyananthan R, Skinner E, Anyaoku V, Richmond W, Sharp P, Johnston DG. The effects of short and long-term growth hormone replacement therapy in hypopituitary adults on lipid metabolism and carbohydrate tolerance. J Clin Endocrinol Metab. 1995 Feb;80(2):356-63. doi: 10.1210/jcem.80.2.7852490.
- [Background] Colao A, di Somma C, Cuocolo A, Spinelli L, Tedesco N, Pivonello R, Bonaduce D, Salvatore M, Lombardi G. Improved cardiovascular risk factors and cardiac performance after 12 months of growth hormone (GH) replacement in young adult patients with GH deficiency. J Clin Endocrinol Metab. 2001 May;86(5):1874-81. doi: 10.1210/jcem.86.5.7464. PMID 11344175
- [Background] Hwu CM, Kwok CF, Lai TY, Shih KC, Lee TS, Hsiao LC, Lee SH, Fang VS, Ho LT. Growth hormone (GH) replacement reduces total body fat and normalizes insulin sensitivity in GH-deficient adults: a report of one-year clinical experience. J Clin Endocrinol Metab. 1997 Oct;82(10):3285-92. doi: 10.1210/jcem.82.10.4311. PMID 9329355
- [Background] Borson-Chazot F, Serusclat A, Kalfallah Y, Ducottet X, Sassolas G, Bernard S, Labrousse F, Pastene J, Sassolas A, Roux Y, Berthezene F. Decrease in carotid intima-media thickness after one year growth hormone (GH) treatment in adults with GH deficiency. J Clin Endocrinol Metab. 1999 Apr;84(4):1329-33. doi: 10.1210/jcem.84.4.5595. PMID 10199774
- [Background] Libby P, Ridker PM. Novel inflammatory markers of coronary risk: theory versus practice. Circulation. 1999 Sep 14;100(11):1148-50. doi: 10.1161/01.cir.100.11.1148. No abstract available. PMID 10484532
- [Background] Ridker PM. Evaluating novel cardiovascular risk factors: can we better predict heart attacks? Ann Intern Med. 1999 Jun 1;130(11):933-7. doi: 10.7326/0003-4819-130-11-199906010-00018. PMID 10375342
- [Background] Ridker PM, Cushman M, Stampfer MJ, Tracy RP, Hennekens CH. Inflammation, aspirin, and the risk of cardiovascular disease in apparently healthy men. N Engl J Med. 1997 Apr 3;336(14):973-9. doi: 10.1056/NEJM199704033361401. PMID 9077376
- [Background] Ridker PM, Buring JE, Shih J, Matias M, Hennekens CH. Prospective study of C-reactive protein and the risk of future cardiovascular events among apparently healthy women. Circulation. 1998 Aug 25;98(8):731-3. doi: 10.1161/01.cir.98.8.731. PMID 9727541
- [Background] Koenig W, Sund M, Frohlich M, Fischer HG, Lowel H, Doring A, Hutchinson WL, Pepys MB. C-Reactive protein, a sensitive marker of inflammation, predicts future risk of coronary heart disease in initially healthy middle-aged men: results from the MONICA (Monitoring Trends and Determinants in Cardiovascular Disease) Augsburg Cohort Study, 1984 to 1992. Circulation. 1999 Jan 19;99(2):237-42. doi: 10.1161/01.cir.99.2.237. PMID 9892589
- [Background] Tracy RP, Lemaitre RN, Psaty BM, Ives DG, Evans RW, Cushman M, Meilahn EN, Kuller LH. Relationship of C-reactive protein to risk of cardiovascular disease in the elderly. Results from the Cardiovascular Health Study and the Rural Health Promotion Project. Arterioscler Thromb Vasc Biol. 1997 Jun;17(6):1121-7. doi: 10.1161/01.atv.17.6.1121. PMID 9194763
- [Background] Kuller LH, Tracy RP, Shaten J, Meilahn EN. Relation of C-reactive protein and coronary heart disease in the MRFIT nested case-control study. Multiple Risk Factor Intervention Trial. Am J Epidemiol. 1996 Sep 15;144(6):537-47. doi: 10.1093/oxfordjournals.aje.a008963. PMID 8797513
- [Background] Ridker PM, Glynn RJ, Hennekens CH. C-reactive protein adds to the predictive value of total and HDL cholesterol in determining risk of first myocardial infarction. Circulation. 1998 May 26;97(20):2007-11. doi: 10.1161/01.cir.97.20.2007. PMID 9610529
- [Background] Fyfe AI, Rothenberg LS, DeBeer FC, Cantor RM, Rotter JI, Lusis AJ. Association between serum amyloid A proteins and coronary artery disease: evidence from two distinct arteriosclerotic processes. Circulation. 1997 Nov 4;96(9):2914-9. doi: 10.1161/01.cir.96.9.2914. PMID 9386157
- [Background] Inoue T, Saito H, Fukushima R, Inaba T, Lin MT, Fukatsu K, Muto T. Growth hormone and insulinlike growth factor I enhance host defense in a murine sepsis model. Arch Surg. 1995 Oct;130(10):1115-22. doi: 10.1001/archsurg.1995.01430100093018. PMID 7575126
- [Background] Geffner M. Effects of growth hormone and insulin-like growth factor I on T- and B-lymphocytes and immune function. Acta Paediatr Suppl. 1997 Nov;423:76-9. doi: 10.1111/j.1651-2227.1997.tb18377.x. PMID 9401546
- [Background] Jarrar D, Wolf SE, Jeschke MG, Ramirez RJ, DebRoy M, Ogle CK, Papaconstaninou J, Herndon DN. Growth hormone attenuates the acute-phase response to thermal injury. Arch Surg. 1997 Nov;132(11):1171-5; discussion 1175-6. doi: 10.1001/archsurg.1997.01430350021003. PMID 9366708
- [Background] Sesmilo G, Biller BM, Llevadot J, Hayden D, Hanson G, Rifai N, Klibanski A. Effects of growth hormone administration on inflammatory and other cardiovascular risk markers in men with growth hormone deficiency. A randomized, controlled clinical trial. Ann Intern Med. 2000 Jul 18;133(2):111-22. doi: 10.7326/0003-4819-133-2-200007180-00010. PMID 10896637
- [Background] Sesmilo G, Miller KK, Hayden D, Klibanski A. Inflammatory cardiovascular risk markers in women with hypopituitarism. J Clin Endocrinol Metab. 2001 Dec;86(12):5774-81. doi: 10.1210/jcem.86.12.8087. PMID 11739438